CLINICAL TRIAL: NCT01556022
Title: Adipose-derived Regenerative Cells in the Treatment of Patients With Chronic Ischemic Heart Disease Not Amenable to Surgical or Interventional Revascularization.
Brief Title: Safety and Feasibility Trial of Adipose-Derived Regenerative Cells in the Treatment of Chronic Myocardial Ischemia
Acronym: ATHENA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: The ATHENA Trial
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Myocardial Ischemia
Keywords: Ischemic heart disease; Coronary artery disease; Chronic heart failure; Cardiovascular disease; Adult stem cells; Adipose derived regenerative cells
MeSH Terms: conditions — Myocardial Ischemia; Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADRCs processed by the Celution System (Experimental): 400,000 adipose-derived regenerative cells (ADRCs) per kilogram (kg) of body weight not to exceed 40,000,000 cells.
  Interventions: Device: ADRCs processed by the Celution System
- Lactated Ringers and Subject's blood (Placebo Comparator): Sterile Lactated Ringers Solution (3mL) mixed with ≤ 0.10 ml of the study Subject's own freshly drawn blood.
  Interventions: Device: Placebo Comparator: Lactated Ringer's and Subject's Blood

INTERVENTIONS:
Device: ADRCs processed by the Celution System — Subjects will undergo liposuction under anesthesia. Lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs. When randomized to ADRCs, intramyocardial injections of ADRCs will be administered via the MYOSTAR injection catheter.
  Other Names: ADRCs; Intramyocardial injections
  Arms: ADRCs processed by the Celution System
Device: Placebo Comparator: Lactated Ringer's and Subject's Blood — Subjects will undergo liposuction under anesthesia. Lipoaspirate will be processed in the Celution System to isolate and concentrate ADRCs. When randomized to Placebo, intramyocardial injections of Placebo will be administered via the MYOSTAR injection catheter.
  Other Names: Placebo
  Arms: Lactated Ringers and Subject's blood

SUMMARY:
This is a prospective, randomized, placebo-controlled, double blind safety and feasibility clinical trial.

DETAILED DESCRIPTION:
To assess the safety and feasibility of Adipose-Derived Regenerative Cells (ADRCs) delivered via an intramyocardial route in the treatment of chronic ischemic heart disease in patients who are not eligible for percutaneous or surgical revascularization.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females 20-80 years of age
2. Significant multi-vessel coronary artery disease not amenable to percutaneous or surgical revascularization in the target area
3. CCS Angina Functional Class II-IV and/or NYHA Stages of Heart Failure Class II or III
4. On maximal medical therapy for anginal symptoms and or heart failure symptoms
5. Hemodynamic stability (Systolic Blood Pressure ≥ 90 mm/Hg, Heart Rate < 110; Pulse-Oxygen > 95)
6. Ejection fraction ≤ 45
7. Left ventricular wall thickness ≥ 8 mm at the target site for cell injection, confirmed by 2D contrast echo within 4 weeks prior to enrollment, free of thrombus

Key Exclusion Criteria:

1. Atrial fibrillation or flutter without a pace maker that guarantees a stable heart rate
2. Unstable angina
3. LV thrombus, as documented by echocardiography
4. Planned staged treatment of CAD or other intervention on the heart
5. Platelet count < 100,000/mm3
6. WBC < 2,000/mm3
7. TIA or stroke within 90 days prior to randomization
8. ICD shock within 30 days of randomization
9. Any condition requiring immunosuppressive medication
10. A high-risk acute coronary syndrome (ACS) or a myocardial infarction within 60 days prior to randomization
11. Revascularization within 60 days prior to randomization
12. Inability to walk on a treadmill except for class IV angina patients who will be evaluated separately
13. Hepatic dysfunction, as defined as aspartate aminotransferase (AST) and /or alanine aminotransferase (ALT) > 1.5 times the upper limit of normal range (x ULN) prior to randomization

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2012-06; Primary Completion 2015-08 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Treatment emergent serious adverse events (SAEs), major adverse cardiac events (MACE), arrhythmia assessment, change in cardiac function and symptoms, and resource utilization | 6 and 12 Months
  Safety endpoints include:
  1. Treatment emergent SAEs
  2. Arrhythmia assessment via Holter monitoring
  3. MACE defined as cardiac death and hospitalization for heart failure
  Feasibility endpoints include:
  1. Change in mVO2 at 6 months
  2. Change in LVESV/LVEDV at 6 months
  3. Change in ejection fraction at 6 months
  4. Change in perfusion defect at 6 months
  5. Resource utilization
  6. Change in heart failure symptoms, angina, and quality of life through 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emerson Perin, MD, PhD, Principal Investigator — Texas Heart Institute, Houston, TX; Timothy Henry, MD, Principal Investigator — Minneapolis Heart Institute Foundation, Minneapolis, MN
Locations (8):
- United States (8):
  - Cardiology, P.C., Birmingham, Alabama
  - Scripps Clinic - Torrey Pines, Scripps Green Hospital, La Jolla, California
  - University of Florida, Gainesville, Florida
  - Florida Hospital-Pepin Heart Institute, Tampa, Florida
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Duke University Hospital, Durham, North Carolina
  - Texas Heart Institute, Houston, Texas
  - University of Utah Health Care, Salt Lake City, Utah

REFERENCES:
- [Result] Henry TD, Pepine CJ, Lambert CR, Traverse JH, Schatz R, Costa M, Povsic TJ, David Anderson R, Willerson JT, Kesten S, Perin EC. The Athena trials: Autologous adipose-derived regenerative cells for refractory chronic myocardial ischemia with left ventricular dysfunction. Catheter Cardiovasc Interv. 2017 Feb 1;89(2):169-177. doi: 10.1002/ccd.26601. Epub 2016 Sep 23. PMID 27148802